CLINICAL TRIAL: NCT06026098
Title: A Prospective Evaluation of Impact of AI Assistance on Workload Associated With Preparation of Rare Tumor Case Reports
Brief Title: Evaluation of Impact of AI Assistance on Workload Associated w Preparation of Rare Tumor Case Repts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-1262
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Burden; Cognitive Symptom
Keywords: artificial intelligence; case report
MeSH Terms: conditions — Neurobehavioral Manifestations | interventions — Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Report with Artificial Intelligence (Experimental): Medical students, resident physicians, or attending physicians report rare cases with using Artificial Intelligence.
  Interventions: Behavioral: Artificial Intelligence
- Case Report without Artificial Intelligence (No Intervention): Medical students, resident physicians, or attending physicians report rare cases without using Artificial Intelligence.

INTERVENTIONS:
Behavioral: Artificial Intelligence — Participants will use the Artificial Intelligence assistance tool for case reports.
  Arms: Case Report with Artificial Intelligence

SUMMARY:
The goal of this study is to explore cognitive burden perceptions among physicians in relation to case report writing. Furthermore, this study evaluates the use of artificial intelligence (AI) assistance as a tool to reduce cognitive burden among providers preparing and submitting case reports. If an AI-tool is helpful in this setting, it may potentially help increase reporting of rare medical events and thereby improve the evidence base for care of these patient populations. This study will occur at a single time point which is expected to last approximately 2 hours. This session will include reviewing two rare tumor cases and then writing a clinical vignette with and without AI assistance.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a physician, medical student, or postdoctoral student.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Subjective Cognitive workload (CWL) | Baseline to 2 hours
  Subjective Cognitive workload (CWL) will be measured while interviews using The National Aeronautics and Space Administration task load (NASA TLX) index is a tool for measuring and conducting a subjective mental workload (MWL) assessment.
  The NASA-TLX is a subjective measure of CWL and is used across many disciplines. The NASA-TLX considers six dimensions-Mental, Physical, and Temporal Demands, Frustration, Effort, and Performance. NASA-TLX scores ≥55 have been associated with reduced performance in numerous settings. NASA-TLX is considered to be the most used subjective measure of CWL. The validated two-stage process with participants performing 15 separate pair-wise comparisons between 6 dimensions of NASA-TLX will be used. A workload score will be marked from low and high for each dimension.
  Score values from 0 -100. The Interpretation Score of NASA TLX for Low 0-9, Medium 10-29, Somewhat high 30-49, High 50-79, and Very high 80-100
Perceived cognitive load | Baseline to 2 hours
  The perceived cognitive load will be measured using System Usability Scale (SUS).
  SUS is a validated post-test questionnaire that measures user satisfaction. Further, studies confirm that SUS is predictive of the impacts of changes to the user interface on usability when multiple changes to a single product were made over a large number of iterations.
  SUS is composed of 10 questions- five positive and five negative statements, each having a five-point scale that ranges from strongly disagree to strongly agree. SUS provides a score (range, 0-100) based on the participant's rating of 10 statements regarding usability with higher scores indicating greater satisfaction with usability.

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Sud, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials